CLINICAL TRIAL: NCT00507130
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled,Dose-Escalation Study to Evaluate the Safety and Tolerability of Multiple-Dose Subcutaneous Administration of MEDI-528, A Humanized Anti-Interleukin-9 Monoclonal Antibody,When Administered to Adults With Mild Persistent Asthma
Brief Title: A Study to Evaluate the Safety and Tolerability of the Administration of MEDI-528 When Administered in Multiple Doses to Adults With Mild Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP131; NCT00507130 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — enokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MEDI528 0.3 mg/kg (Experimental): MEDI-528 at a dose of 0.3 mg/kg administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Interventions: Biological: MEDI528 0.3 mg/kg
- MEDI528 1 mg/kg (Experimental): MEDI-528 at a dose of 1 mg/kg administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Interventions: Biological: MEDI528 1 mg/kg
- MEDI528 3 mg/kg (Experimental): MEDI-528 at a dose of 3 mg/kg administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Interventions: Biological: MEDI528 3 mg/kg
- PLACEBO (Placebo Comparator): Placebo administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Interventions: Other: PLACEBO

INTERVENTIONS:
Biological: MEDI528 0.3 mg/kg — MEDI-528 at a dose of 0.3 mg/kg administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Arms: MEDI528 0.3 mg/kg
Biological: MEDI528 1 mg/kg — MEDI-528 at a dose of 1 mg/kg administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Arms: MEDI528 1 mg/kg
Biological: MEDI528 3 mg/kg — MEDI-528 at a dose of 3 mg/kg administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Arms: MEDI528 3 mg/kg
Other: PLACEBO — Placebo administered twice weekly as a subcutaneous (SC) dose for 4 weeks
  Arms: PLACEBO

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of escalating multiple SC doses of MEDI-528 in adult patients with mild persistent asthma.

DETAILED DESCRIPTION:
The secondary objectives of this study are to:

1. Assess the PK of MEDI-528; and
2. Assess the IM of MEDI-528 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, age 18 through 65 years of age at time of screening;
* Weight ≤ 100 kg and body mass index ≤ 35;
* Written informed consent obtained from the patient prior to receipt of any study medication or beginning study procedures;
* Previously documented diagnosis of asthma based on episodic symptoms of airflow obstruction such as wheezing or chest tightness, with alternative diagnoses (e.g., chronic obstructive pulmonary disease) ruled out;
* Currently receiving treatment with short-acting β2 agonists, ICS at doses ≤ 264 μg/day fluticasone or equivalent, or both (National Heart, Lung, and Blood Institute [NHLBI], 2002);
* FEV1 or peak expiratory flow (PEF) ≥ 80% of predictable value;
* Have had a diagnosis of mild persistent asthma, defined as having asthma symptoms with a frequency of more than twice a week but less than once daily, or nighttime symptoms with a frequency of more than twice a month but less than once a week (NHLBI, 2002);
* Have AHR based on documented clinical history of either methacholine inhalation challenge with PC20 ≤ 16 mg/mL or partial reversibility of ≤ 12% in FEV1 within the past 18 months (including screening);
* Able to provide spirometry readings that meet American Thoracic Society/European Respiratory Society standards (Miller, 2005);
* Sexually active females, unless surgically sterile or at least 1 year post-menopausal, must use an effective method of avoiding pregnancy (including oral, implanted, or transdermal contraceptives, intrauterine device, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 21 days prior to the first dose of study drug, and must agree to continue using such precautions through Study Day 150. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active males, unless surgically sterile, must likewise use an effective method of birth control (condom) and must agree to continue using such precautions through Study Day 150;
* Ability to complete the study period, including follow-up period, of up to 150 days; and
* Willing to forego other forms of experimental treatment and study procedures during the study.

Exclusion Criteria:

* Receipt of MEDI-528 in any previous clinical study or prior randomization into the trial;
* History of allergy or reaction to any component of the MEDI-528 formulation;
* Lung disease other than persistent asthma (e.g. chronic bronchitis);
* FEV1 < 80% of predicted values;
* History of severe asthma or asthma exacerbation requiring intubation;
* Use of systemic immunosuppressive drugs including systemic corticosteroids or ICS with doses > 264 μg/day fluticasone or equivalent within 4 weeks prior to Study Day 0;
* Use of long-acting β2 agonists, theophylline, cromolyn sodium, nedocromil sodium, leukotriene receptor antagonists, or any other inhaled or systemic medication for asthma (except short-acting β2 agonists or ICS at doses ≤ 264 μg/day fluticasone or equivalent) within the 2 weeks prior to Study Day 0;
* Current use of any β-adrenergic antagonist (e.g., propranolol);
* Any disease or illness, other than asthma, that may require the use of systemic corticosteroids during the study period;
* Acute illnesses or evidence of significant active infection, such as fever ≥ 38.0°C (100.5°F) at screening and up through time of the first dose of study drug;
* Current allergy vaccination therapy (desensitization immunotherapy), with less than 3 months of stable maintenance doses prior to screening;
* Receipt of any investigational drug therapy within 30 days or any biologic(s) within 5 half-lives of the agent prior to the first dose of study drug through Study Day 150;
* Receipt of any therapy with a leukocyte-depleting agent unless recovery in white cell count has been documented before screening;
* Pregnancy (sexually active females must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to study drug administration on Study Day 0);
* Lactating or breastfeeding woman;
* Evidence of infection with hepatitis B or C virus, or human immunodeficiency virus-1 or -2 (HIV-1 or HIV-2), or active infection with hepatitis A;
* History of significant systemic disease (e.g., cancer, infection, hematological, renal, hepatic, coronary artery disease or other cardiovascular disease, endocrinologic, neurologic, rheumatologic, or gastrointestinal disease);
* History of cancer other than non-melanoma skin cancer or cervical carcinoma-in-situ treated with apparent success with curative therapy (remission for ≥ 1 year prior to screening);
* History of primary immunodeficiency;
* History of pancreatitis;
* History of use of tobacco products of more than one cigarette per month or equivalent within 1 year prior to randomization or history of smoking of ≥ 10 pack-years;
* Elective surgery planned during the study period through Study Day 150;
* Clinically significant abnormalities on physical examination (other than asthma) prior to the first dose of study drug (including but not limited to splenomegaly); Clinically significant abnormality, as determined by the investigator, on 12-lead ECG, MRI, or chest radiograph at the time of screening;
* At the time of screening, any abnormality of the following measurements: hemoglobin, total white blood cell count (WBC), platelet count, aspartate transaminase (AST), alanine transaminase (ALT), amylase, or serum creatinine above the upper limits of normal (ULN); or other abnormal laboratory values in the screening panel that, in the opinion of the principal investigator, are judged to be clinically significant;
* Evidence of any systemic disease or respiratory disease (other than asthma), any finding upon physical examination or history of any disease that, in the opinion of the investigator or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study; or
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or family members of such individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Parker, M.D., Study Director — MedImmune LLC
Locations (9):
- United States (6):
  - Colorado Allergy & Asthma Centers, PC, Denver, Colorado
  - Northeast Medical Research Associates, Inc., North Dartmouth, Massachusetts
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Spartanburg Medical Research, Spartanburg, South Carolina
- Canada (3):
  - McMaster University, Hamilton, Ontario
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Hopital Laval, Québec, Quebec

REFERENCES:
- [Derived] Parker JM, Oh CK, LaForce C, Miller SD, Pearlman DS, Le C, Robbie GJ, White WI, White B, Molfino NA; MEDI-528 Clinical Trials Group. Safety profile and clinical activity of multiple subcutaneous doses of MEDI-528, a humanized anti-interleukin-9 monoclonal antibody, in two randomized phase 2a studies in subjects with asthma. BMC Pulm Med. 2011 Feb 28;11:14. doi: 10.1186/1471-2466-11-14. PMID 21356110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 subjects were entered into the study between 28Jun2007 and 17Jul2008 at 8 sites in the United States of America (5 sites) and Canada (3 sites).
Pre-assignment Details: Treatment assignments were determined using a block randomization procedure at a 3:1 active treatment-to-placebo ratio through an interactive voice response system (IVRS). When a subject was assigned a Participant Identification Number by the IVRS, the subject was considered randomized into the study.
Groups:
- MEDI528 0.3 mg/kg: MEDI-528 at a dose of 0.3 mg/kg administered twice weekly as a SC dose for 4 weeks
- MEDI528 1 mg/kg: MEDI-528 at a dose of 1 mg/kg administered twice weekly as a SC dose for 4 weeks
- MEDI528 3 mg/kg: MEDI-528 at a dose of 3 mg/kg administered twice weekly as a SC dose for 4 weeks
Period: Overall Study
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Started | 9 | 9 | 9 | 9
Completed | 8 | 9 | 8 | 8
Not Completed | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — SERIOUS EVENT OF ASTHMA EXACERBATION | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (13.2) | 38.2 (16.3) | 33.2 (11.9) | 28.9 (10.7) | 34.7 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 5 | 5 | 26
  Male | 1 | 1 | 4 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Number of participants experiencing adverse events (includes both adverse events and serious adverse events)
Time Frame: Days 0 - 150
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 9 | 9 | 9 | 9

2. Primary Outcome: Incidence of Abnormal Troponin Levels
Description: Number of participants with troponin levels greater than upper limit of normal
Time Frame: Days 0, 14, 28, 56, 84, and 150
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 1

3. Primary Outcome: Incidence of Abnormal Clinically Significant Electrocardiogram (ECG) Results
Description: Number of participants with abnormal clinically significant ECG results
Time Frame: Days -14 to -1, 14, 28, 56, 84, and 150
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Incidence of Abnormal Clinically Significant Magnetic Resonance Imaging (MRI) Results
Description: Number of participants experiencing abnormal clinically significant MRI results
Time Frame: Days -14 to -1 and 28
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of participants experiencing serious adverse events
Time Frame: Days 0 - 150
Population: All subjects who received at least one dose of investigational product (MEDI-528 or placebo)
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 1 | 0 | 0 | 0

6. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) to MEDI-528
Description: Number of participants with ADA to MEDI-528
Time Frame: Days 0, 28, 56, 84, 119, and 150
Population: All subjects who received at least one dose of MEDI-528
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Time to Observed Maximum Serum Concentration (Tmax)
Description: Tmax of MEDI-528
Time Frame: Days 0, 3, 7, 10, 14, 17, 21, 24, 26, 28, 31, 35, 42, 49, 56, 70, 84, 119, and 150
Population: All subjects who received at least one dose of MEDI-528 and had blood samples analyzed for pharmacokinetic analysis
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 0 | 8 | 9 | 9
Day |  | 3.5 (2.1) | 3.7 (2.3) | 3.9 (2.6)

8. Secondary Outcome: Observed Maximum Serum Concentration (Cmax)
Description: Cmax of MEDI-528
Time Frame: Days 0, 3, 7, 10, 14, 17, 21, 24, 26, 28, 31, 35, 42, 49, 56, 70, 84, 119, and 150
Population: All subjects who received at least one dose of MEDI-528 and had blood samples analyzed for pharmacokinetic analysis
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 0 | 8 | 9 | 9
Micrograms per milliliter |  | 13.7 (2.7) | 52.1 (33.0) | 105.5 (31.0)

9. Secondary Outcome: Terminal Phase Half-life (T1/2)
Description: T1/2 of MEDI-528
Time Frame: Days 0, 3, 7, 10, 14, 17, 21, 24, 26, 28, 31, 35, 42, 49, 56, 70, 84, 119, and 150
Population: All subjects who received at least one dose of MEDI-528 and had blood samples analyzed for pharmacokinetic analysis
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Number analyzed (Participants) | 0 | 8 | 9 | 9
Day |  | 37.1 (7.5) | 35 (11.5) | 37.7 (7.5)

ADVERSE EVENTS:
Arm/Group | PLACEBO | MEDI528 0.3 mg/kg | MEDI528 1 mg/kg | MEDI528 3 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=9) | MEDI528 0.3 mg/kg (N=9) | MEDI528 1 mg/kg (N=9) | MEDI528 3 mg/kg (N=9)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=9) | MEDI528 0.3 mg/kg (N=9) | MEDI528 1 mg/kg (N=9) | MEDI528 3 mg/kg (N=9)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (8)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 3 (4) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (2) | 1 (2) | 2 (2) | 3 (5)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood chloride decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood chloride increased (Investigations) | 2 (2) | 1 (3) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 3 (3) | 5 (8) | 3 (5) | 1 (3)
Blood potassium decreased (Investigations) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
False positive laboratory result (Investigations) | 4 (7) | 2 (3) | 1 (3) | 4 (6)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (5) | 1 (2)
White blood cell count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.